CLINICAL TRIAL: NCT03776799
Title: BEST SFA Pilot Study - Best Endovascular STrategy for Complex Lesions of the Superficial Femoral Artery Comparing a Stent-avoiding (study Arm) Versus Stent-preferred (control Arm) Approach Within a Prospective, Randomized, Multi-center Trial
Brief Title: BEST SFA Pilot Study - Best Endovascular STrategy for Complex Lesions of the Superficial Femoral Artery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Dierk Scheinert, Clinic director, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP_18/001
Record Dates: First submitted 2018-12-05; First posted 2018-12-17 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stent-avoiding approach (Other): using clinically proven drug coated balloons
  Interventions: Device: Stent-avoiding
- Stent-based approach (Other): using drug eluting nitinol stents. Interwoven nitinol stents in heavily calcified lesions at the operator's discretion.
  Interventions: Device: Stent-based

INTERVENTIONS:
Device: Stent-avoiding — Percutaneous transluminal angioplasty (PTA), in which a balloon is advanced and inflated in the obstructed artery for several seconds to minutes, has become the standard endovascular treatment for peripheral arteries
  Arms: Stent-avoiding approach
Device: Stent-based — Stenting, in which a stent is advanced and implanted in the obstructed artery, has become the standard endovascular treatment for peripheral arteries
  Arms: Stent-based approach

SUMMARY:
Prospective, multi-center 1:1 randomized trial to compare efficacy and safety of a stent-avoiding (using drug coated balloons) versus a stent-preferred (using drug eluting or interwoven stents) approach for treatment of complex femoropopliteal lesions TASC II (TransAtlantic Inter-Society Consensus for the Management of Peripheral Arterial Disease) Type B-D (stenosis >10cm, occlusions >5cm).

DETAILED DESCRIPTION:
Prospective, multi-center 1:1 randomized Study.

Patients will be stratified according to a stent-avoiding (study arm) or stent-preferred (control arm)

In total 120 patient will be enrolled in this study, each strata will include 60 patients.

All enrolled patients will be followed up for 24 month to asses the incidence of restenosis by duplex ultrasound and major adverse events.

Follow-up visits occur at 6, 12 and 24 month intervals as well as telephone visit after 1,36, 48 and 60 month.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≥ 18
2. Subject has been informed of the nature of the study, agrees to participate, and has signed a Medical Ethics Committee approved consent form Subject understands the duration of the study, agrees to attend follow-up visits, and agrees to complete the required testing.
3. Subject has a de novo or restenotic lesion with ≥ 70% stenosis documented angiographically and no prior stent in the target lesion.
4. Rutherford Becker Classification 2-4
5. Both treatment options seem feasible at the operator's discretion
6. Femoropopliteal lesions classified as TASC II Type B-D with a maximum lesion length ≤ 30cm not involving the infrageniculate popliteal artery are eligible.
7. Reference vessel diameter (RVD) ≥ 4 mm and ≤ 6.5 mm by visual estimation.
8. Patency of at least one (1) infrapopliteal artery to the ankle (< 50% diameter stenosis) in continuity with the native femoropopliteal artery. The inflow artery(ies) cannot be treated using a drug eluting stent or drug coated balloon
9. A guidewire has successfully traversed the target treatment segment.

Exclusion Criteria:

1. Failure to successfully cross the target lesion
2. Angiographic evidence of severe calcification that makes a stent-avoiding approach not feasible at the operator's discretion.
3. Femoropopliteal lesions classified as TASC II Typ A (single stenosis >=10cm and single occlusion >=5cm)
4. Presence of fresh thrombus in the lesion.
5. Presence of aneurysm in the target vessel/s
6. Presence of a stent in the target lesion
7. Prior vascular surgery of the target lesion.
8. Stroke or heart attack within 3 months prior to enrollment
9. Any planned surgical procedure or intervention performed within 30 days prior to or post index procedure
10. SFA or PPA disease in the opposite leg that requires treatment at the index procedure
11. Enrolled in another investigational drug, device or biologic study that interferes with the study
12. Life expectancy of less than one year
13. Known allergies or sensitivity to heparin, aspirin, other anticoagulant/ antiplatelet therapies, paclitaxel or contrast media that cannot be adequately pre-treated prior to index procedure
14. Rutherford classification of 0, 1, 5 or 6.
15. Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy.
16. Platelet count <100,000 mm3 or >600,000 mm3
17. Receiving dialysis or immunosuppressant therapy
18. Pregnant or lactating females.
19. History of major amputation in the same limb as the target lesion
20. Chronic kidney disease (serum creatinine > 3 mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Primary patency - Absence of clinically-driven target lesion revascularization (CD-TLR) and/or restenosis defined as a peak systolic velocity ratio (PSVR) > 2.4 assessed by ultrasound | 1 Year

SECONDARY OUTCOMES:
Walking capacity - Walking capacity assessed by Walking impairment questionnaire score at 6, 12 and 24 | 2 Year
  The graded score is multiplied by a pre-specified weight for each distance, speed, or number of stair flights. The products are summed and divided by the maximum possible score to obtain a percent score, ranging from 0 (representing the inability to perform any of the tasks) to 100 (representing no difficult with any of the tasks)
Ankle-brachial index - Clinical improvment assessed by Ankle-brachial index at 6, 12 and 24 month | 2 Year
  The ABI is calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressure in the arm. An ABI between and including 0.9 and 1.2 considered normal (free from significant PAD), while a lesser than 0.9 indicates arterial disease
Rutherford category - Clinical improvment assessed by Rutherford category at 6, 12 and 24 month | 2 Year
  This classification system consists of four grades and seven categories (categories 0-6):
  Grade 0, Category 0: asymptomatic Grade I, Category 1: mild claudication Grade I, Category 2: moderate claudication Grade I, Category 3: severe claudication Grade II, Category 4: rest pain Grade III, Category 5: minor tissue loss; ischemic ulceration not exceeding ulcer of the digits of the foot Grade IV, Category 6: major tissue loss; severe ischemic ulcers or frank gangrene
Freedom from device and procedure-related death, all-cause death, target limb major amputation and clinically-driven target lesion revascularization | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, Prof. Dr., Principal Investigator — University Clinic Leipzig
Locations (1):
- University Clinic Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wittig T, Schmidt A, Fuss T, Thieme M, Maiwald L, Dusing S, Konert M, Fischer A, Scheinert D, Steiner S. Randomized Trial Comparing a Stent-Avoiding With a Stent-Preferred Strategy in Complex Femoropopliteal Lesions. JACC Cardiovasc Interv. 2024 May 13;17(9):1134-1144. doi: 10.1016/j.jcin.2024.03.015. PMID 38749594